CLINICAL TRIAL: NCT06629740
Title: A Post-market Clinical Follow-up Investigation in Healthy Volunteers Measuring Eye Parameters to Verify Performance and Safety of Previct® Drugs for Monitoring of Patients in Treatment of Substance Use Disorder
Brief Title: A Study of a Mobile Phone Application Measuring the Eyes Before and After Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kontigo Care AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCClin03; NL87202.058.24 (Other: Central Committee on Research Involving Human Subjects (CCMO), Netherlands)
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Substance Use Disorder (SUD)
Keywords: substance use disorder; post-market clinical follow-up; eye monitoring; smartphone; app
MeSH Terms: conditions — Substance-Related Disorders; Alzheimer Disease | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of two arms for deciding upon which of the two medicines (phenethylamine or cannabinoid) to be administered through a single application at visit 2. The randomization will also take into account which one of three different smartphone brands with the Previct Drugs mobile phone application preinstalled to be used by the subject during the study.
  The study aims to enroll 30 subjects, 12 subjects in the phenethylamine group and 18 subjects in the cannabinoid group. The dropout rate is estimated to 10%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabinoid (Experimental): A single administration of cannabinoid where a CE-marked eHealth system will be used before and after intake.
  Interventions: Device: Measurements with a eHealth system
- Phenethylamine (Experimental): A single administration of phenethylamine where a CE-marked eHealth system will be used before and after intake.
  Interventions: Device: Measurements with a eHealth system

INTERVENTIONS:
Device: Measurements with a eHealth system — The eHealth system Previct Drugs is a CE marked medical device intended to be used in treatment of substance use disorder (SUD) to support and monitor patients' treatment. Previct Drugs consists of a mobile phone application used to perform self-administered eye-scanning, a web-based careportal used by the caregiver, a database for storage, handling, and analysis of reported data, and an admin portal for the manufacturer to register and administer customers. In this study, Previct Drugs will be used by healthy volunteers for performing measurements before and after intake of a commonly used medicine to simulate drug intake.

SUMMARY:
This is a post-market clinical follow-up study on an approved CE-marked eHealth system where a mobile phone application is used to measure the pupils and eye measurements to monitor the use of different drug substances. The goal of the study is to collect additional information when using the system and to improve the current models for indicating the use of cannabinoids and phenethylamines.

Drug intake of cannabinoid or phenethylamine will in this study be simulated using two commonly used medicines.

The study will include healthy volunteers where each participant will participate in the study for approximately 10 days. The participant will be using the mobile phone application for about a week, first at the clinic and then in the home environment. After approximately a week the participant will visit the clinic to be administered with the selected medicine whereafter the mobile phone application will be used for up to 5 hours. A final phone call will be taken place at approximately day 10, whereafter the participant has completed the study.

DETAILED DESCRIPTION:
This is a controlled, prospective, post-market clinical follow-up study that aims to collect additional data on performance and safety of the CE-marked eHeatlh system Previct Drugs. Previct Drugs is intended to be used in treatment of substance use disorder (SUD) to support and monitor patients' treatment. The system relies on self-administered eye scanning performed with a mobile phone application where the analysis of the eye´s reaction on intake of drug substances gives an indication of different drug substances. The clinical data collected in this study is an important step to verify and improve the algorithms of Previct Drugs, and to improve the mathematical models for indicating the use of the substances cannabinoids and phenethylamines.

Drug intake will in this study be simulated by a controlled single application of commonly used medicines from cannabinoids and phenethylamine.

The study will enroll and follow 30 male and female healthy volunteers for participation of approximately 10 days. The study will consist of two visits to the clinic, and one follow-up telephone call before the participant has completed the study. Baseline data will be collected at the first visit on Day 0, including usage of Previct Drugs, followed by usage of Previct Drugs in the home environment for about one week. At visit 2 on Day 7, the subject will be administered with the medicine he/she has been randomized to and thereafter use Previct Drugs for up to 5 hours. A final follow-up telephone call will take place approximately at day 10 before the participant has completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteers.
2. Age 18 to 55 years.
3. BMI between 18.5-30 kg/m2.
4. Weight between 50-100 kg.
5. Healthy as determined by the investigator or designee based on pre-investigational medical and surgical history, and health examination at enrollment.
6. Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to enrollment) must have a negative urine pregnancy test at enrollment and at visit 2 and must agree to use a medically acceptable contraception from enrollment until clinical investigation completion.
7. No current drug usage defined as a negative urine drug test at enrollment and at visit 2.
8. Able to use Previct Drugs after initial training (defined as successfully performing a test set after trying maximum three times per measurement).
9. Voluntarily agrees to participate and has duly singed the Informed Consent Form.

Exclusion Criteria:

1. Participating in another clinical investigation which may affect the clinical investigation outcome according to clinical judgement.
2. Previously participated in the KCClin01 investigation.
3. Pregnant or lactating.
4. Blind and/or deaf.
5. Clinically abnormal ECG, according to the investigator. QTcF time above 450 ms at enrollment.
6. Resting heart rate above 90 BPM.
7. Current or recent history of alcohol misuse assessed by AUDIT where ≥6 points for women or ≥8 points for men indicates a potential misuse.
8. Current or history of psychiatric disorder or drug misuse assessed by M.I.N.I where the outcome will be based on clinical judgement.
9. Any disease or condition that may influence pupillary reflexes based on clinical judgement.
10. Undergone eye surgery that may influence pupillary reflexes based on clinical judgement.
11. Ongoing treatment with medications which may interfere with eye measurements based on clinical judgement.
12. Ongoing treatment with medications which may interfere with any of the medicinal products to be used.
13. History or presence of allergy or serious reaction to the medicinal products to be used.
14. History or presence of cardiovascular disease, e.g., arteriosclerosis, hypertension, or cor pulmonale.
15. History or presence of sleep-related breath disorder.
16. History or presence of gastrointestinal disease, e.g., paralytic ileus, acute abdomen, delayed gastric emptying, or chronic constipation.
17. History or presence of pulmonary disease, e.g., acute pulmonary insufficiency, severe respiratory depression with hypoxia, chronic obstructive lung disease, or bronchial asthma.
18. History or presence of autoimmune neuromuscular disease, e.g., myasthenia gravis.
19. Not able to read or understand the local language.
20. Any other condition that as judged by the investigator may make the follow-up or investigation inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Verify if self-administered eye scanning using a mobile phone application, using native key features (alone or in predefined combination(s)), can indicate use of each medicine (D1-D2). | Day 7 (+/- 2 days)
  For each medicine (D1-D2), changes for each subject in key features (alone or in predefined combination(s)) between baseline at visit 2 and under the influence of D1-D2 at LC-MS/MS defined peak concentration, using native key features.
  Key feature is defined as a predefined characteristic obtained from an eye measurement such as pupil size or motion of iris position over time.

SECONDARY OUTCOMES:
Verify if self-administered eye scanning using a mobile phone application, after refinement of the method for establishing key features (alone or in predefined combination(s)), can indicate the use of each medicine (D1-D2). | Day 7 (+/- 2 days)
  For each medicine (D1-D2), changes for each subject in key features (alone or in predefined combination(s) as described in the primary endpoint), between baseline at visit 2 and under the influence of D1-D2 at LC-MS/MS defined peak concentration, using refined key features.
  Refined key feature is defined as a predefined characteristic obtained from an eye measurement such as pupil size or motion of iris position over time, where underlying algorithms have been refined.
Evaluate the first and last time after medicine intake of D1 or D2 when refined key eye features, alone or in predefined combination(s), differ from baseline. | Day 7 (+/- 2 days)
  For each medicine (D1-D2), changes in refined key features alone or in predefined combination(s), between baseline and under the influence of D1-D2 at 10 min and up to 5 h after medicinal product administration. The comparison is only made using the 5 key features with the lowest p-values from S1.
  Refined key feature is defined as a predefined characteristic obtained from an eye measurement such as pupil size or motion of iris position over time, where underlying algorithms have been refined.
Evaluate the difference between refined drug naïve test data collected at the clinic and compared with tests performed in home environment. | From Day 0 to Day 7 (+ 2 days)
  For each subject, differences between refined key features taken at the clinic (baseline visit 2) and measurements taken in home environment under similar light conditions. This will be performed only with Dbase, Dcon, MCA, MCV. Two different ambient light conditions, as measured with the smartphones, will be compared for dimmed (20-150 Lux) and bright (150-500 Lux) light.
  Refined key feature is defined as a predefined characteristic obtained from an eye measurement such as pupil size, where underlying algorithms have been refined.
Evaluate if the refined drug naïve key features (alone or in predefined combination(s)), collected at baseline differs from data collected at peak plasma concentration under the influence of D1-D2 without compensating for intra-individual variation. | Day 7 (+/- 2 days)
  For each medicine (D1-D2), differences between refined key features (for the 5 key features with lowest p-value as found in S1, or in predefined combination(s)) observed for the cohort collected under the influence of D1-D2 at peak LC-MS/MS defined peak concentration, and observations collected for the cohort when drug naive (baseline visit 2). In this analysis data will be analyzed at group level (drug influenced and drug naive) without using intra-individual changes. (Hence, the groups are handled as two independent cohorts).
  Refined key feature is defined as a predefined characteristics obtained from an eye measurement such as pupil size or motion of iris position over time, where underlying algorithms have been refined.

OTHER OUTCOMES:
Incidence and severity of adverse events. | Throughout the study from enrollment until study completion.
  The incidence and severity of adverse events associated with Previct Drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Markku Hämäläinen, PhD, Study Chair — Kontigo Care AB
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided